CLINICAL TRIAL: NCT06867380
Title: A Feasibility, Prospective, Repeated-measures Investigation to Evaluate Sound Coding Enhancements in Adult Cochlear Implant Recipients: A Master Umbrella Investigation
Brief Title: An Investigation to Evaluate Sound Coding Enhancements in Adult Cochlear Implant Recipients
Acronym: SONORA-MU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AI5838
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-03

CONDITIONS: Cochlear Implant Recipients; Hearing Loss, Cochlear
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Masking Description: Investigational sound coding strategy and default sound coding comparator is blinded to the participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational sound coding strategy/Default sound coding strategy (Sub A) (Experimental): Tested with investigational and default sound coding strategies
  Interventions: Device: Investigational sound coding strategy; Device: Cochlear default sound coding strategy

INTERVENTIONS:
Device: Investigational sound coding strategy — SPARC (Stimulation Place and Rate Coding) sound coding strategies
Device: Cochlear default sound coding strategy — ACE (Advanced Combination Encoder) sound coding strategy

SUMMARY:
This study will evaluate a range of experimental sound coding strategies that may improve hearing for cochlear implant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Users of an approved Nucleus cochlear implant.
* Aged 18 years or older (no upper age limit).
* Open set speech understanding sufficient to complete the study protocol as judged by the investigator.
* Fluent speaker in the language used to assess speech perception performance, as determined by the investigator.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the investigator.
* Additional health factors, known to the investigator, that would prevent or restrict participation in the audiological evaluations.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless the other investigation was/is a Cochlear sponsored investigation and determined by the investigator or Sponsor to not impact this investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Paired difference in Speech Reception Threshold (SRT) score (dB) between the investigational sound coding strategy and the default sound coding strategy | 0 to 12 weeks
  Speech perception in noise will be measured using the Australian Speech Test in Noise (AuSTIN) with speech presented at 65 dB SPL in adaptive 4-talker babble noise, both presented in front of the listener. It is scored as a Speech Reception Threshold (SRT), which reflects the volume of speech signal (in decibels, dB) relative to the background noise required for the subject to achieve 50% correct. For example, a score of 2dB SRT means the subject requires the speech to be 2dB louder than the background noise in order to correctly identify 50% of the target sentence. Range: -30dB to +30dB. Lower scores reflect a better outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - HEARnet Clinical studies, Carlton, Victoria
  - Cochlear Melbourne, East Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No